CLINICAL TRIAL: NCT04837638
Title: Diet Quality and Coronary Artery Calcification in Adults With Heterozygous Familial Hypercholesterolemia
Acronym: FH-CAC
Status: Active, not recruiting | Type: Observational
Sponsor: Laval University (Other)
Collaborators: Centre de Recheche du Centre Hospitalier Université Laval (Other); Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec (Other)
Responsible Party: Principal Investigator, Jean-Philippe Drouin-Chartier, Professor, Laval University
Other Study IDs: FH-CAC (MP-20-2021-5767)
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Hypercholesterolemia, Familial; Calcification; Heart; Diet Habit
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Calcinosis; Feeding Behavior | interventions — Diet

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum and plasma.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with HeFH: Adult men and women aged 18 to 65 years with genetically-defined HeFH.
  Interventions: Behavioral: Diet

INTERVENTIONS:
Behavioral: Diet — No intervention. Cross-section assessment of the relationship between diet, medication, lifestyle and coronary artery calcification.

SUMMARY:
The overarching objective is to evaluate the relationship between diet and coronary artery calcification in patients with heterozygous familial hypercholesterolemia (HeFH). We will recruit adults with HeFH. They will have to complete questionnaires on diet, medication and lifestyle. Coronary artery calcification will be measured in each patient using a CT scan. Physiological and biochemical data will be collected.

DETAILED DESCRIPTION:
The proposed research will deploy as cross-sectional study including treated adults with genetically-defined HeFH. Once recruited, participants will be asked to complete web-based questionnaires on diet, medication and lifestyle. They will thereafter complete a clinical assessment at the Clinical Investigation Unit of the NUTRISS-INAF Research Centre. Study staff will measure participants' height, weight, and waist circumference. Participants' blood pressure will be measured using an automatic blood pressure monitor (BP Thru, Omron) after sitting quietly for 10 minutes. Three sequential readings will be taken with three minutes between readings. Fasting blood samples (10 mL) will be collected from an antecubital vein. Body composition will be assessed with dual-energy X-ray absorptiometry (DEXA). Finally, participants will be asked to provide the full list of medication they are using, including type, dose and duration of use. Later on the same day, participants will undergo the non-contrast CT scan at the Quebec Heart and Lung Institute. Multidetector CT scans without contrast will be performed using a 256 slices helical scanner (Brilliance iCT, Philips).

ELIGIBILITY:
Inclusion Criteria:

- Genetically-defined heterozygous familial hypercholesterolemia

Exclusion criteria:

* Homozygous FH
* Personal history of cardiovascular disease
* Personal history of cancer

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult men and women with genetically-defined HeFH
Sampling Method: Non-Probability Sample
Enrollment: 258 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Relationship between diet quality and coronary artery calcification (CAC) | Diet questionnaire completion and CAC measurement will be completed with a 3 weeks period.
  Diet quality indices reflecting different dimensions of diet will be used as the main exposure, including the Alternative Mediterranean Diet Index (AMED, 9-45 points), the Alternative Healthy Eating Index (AHEI, 0-100 points), the Dietary Approach to Stop Hypertension index (DASHi, 8-40 points), the healthy plant-based diet index (hPDI, 18-90 points) and the unhealthy plant-based diet index (uPDI, 18-90 points). Higher scores reflect higher diet quality, except for the uPDI which reflect lower diet quality. CAC will be measured using non-constrat CT scan. CAC scores will be quantified with the Agatston scoring method. Higher CAC scores reflect higher CAC.

SECONDARY OUTCOMES:
Relationship between diet quality and LDL-cholesterol. | Diet questionnaire completion and CVD risk factor measurement will be completed with a 3 weeks period.
  Diet quality indices reflecting different dimensions of diet will be used as the main exposure, including the Alternative Mediterranean Diet Index (AMED, 9-45 points), the Alternative Healthy Eating Index (AHEI, 0-100 points), the Dietary Approach to Stop Hypertension index (DASHi, 8-40 points), the healthy plant-based diet index (hPDI, 18-90 points) and the unhealthy plant-based diet index (uPDI, 18-90 points). Higher scores reflect higher diet quality, except for the uPDI which reflect lower diet quality. LDL-cholesterol will be measured using standard procedures from the fasting blood sample collected on the same day of the CT-scan.
Relationship between diet quality and Lipoprotein (a). | Diet questionnaire completion and CVD risk factor measurement will be completed with a 3 weeks period.
  Diet quality indices reflecting different dimensions of diet will be used as the main exposure, including the Alternative Mediterranean Diet Index (AMED, 9-45 points), the Alternative Healthy Eating Index (AHEI, 0-100 points), the Dietary Approach to Stop Hypertension index (DASHi, 8-40 points), the healthy plant-based diet index (hPDI, 18-90 points) and the unhealthy plant-based diet index (uPDI, 18-90 points). Higher scores reflect higher diet quality, except for the uPDI which reflect lower diet quality. Lipoprotein (a) will be measured using standard procedures from the fasting blood sample collected on the same day of the CT-scan.
Relationship between diet quality and intuitive eating. | Diet questionnaire completion and psychological aspects of eating measurement will be completed with a 3 weeks period.
  Diet quality indices reflecting different dimensions of diet will be used as the main exposure, including the Alternative Mediterranean Diet Index (AMED, 9-45 points), the Alternative Healthy Eating Index (AHEI, 0-100 points), the Dietary Approach to Stop Hypertension index (DASHi, 8-40 points), the healthy plant-based diet index (hPDI, 18-90 points) and the unhealthy plant-based diet index (uPDI, 18-90 points). Higher scores reflect higher diet quality, except for the uPDI which reflect lower diet quality. Intuitive eating will be measured using the Intuitive Eating Scale.
Relationship between diet quality and physical activity | Diet questionnaire completion and lifestyle habit measurement will be completed with a 3 weeks period.
  Diet quality indices reflecting different dimensions of diet will be used as the main exposure, including the Alternative Mediterranean Diet Index (AMED, 9-45 points), the Alternative Healthy Eating Index (AHEI, 0-100 points), the Dietary Approach to Stop Hypertension index (DASHi, 8-40 points), the healthy plant-based diet index (hPDI, 18-90 points) and the unhealthy plant-based diet index (uPDI, 18-90 points). Physical activity will be assessed using the Godin physical activity questionnaire.
Relationship between diet quality and sleep. | Diet questionnaire completion and lifestyle habit measurement will be completed with a 3 weeks period.
  Diet quality indices reflecting different dimensions of diet will be used as the main exposure, including the Alternative Mediterranean Diet Index (AMED, 9-45 points), the Alternative Healthy Eating Index (AHEI, 0-100 points), the Dietary Approach to Stop Hypertension index (DASHi, 8-40 points), the healthy plant-based diet index (hPDI, 18-90 points) and the unhealthy plant-based diet index (uPDI, 18-90 points). Sleep will be assessed using the Pittsburgh Sleep Quality Index.
Relationship between diet quality and substance use. | Diet questionnaire completion and lifestyle habit measurement will be completed with a 3 weeks period.
  Diet quality indices reflecting different dimensions of diet will be used as the main exposure, including the Alternative Mediterranean Diet Index (AMED, 9-45 points), the Alternative Healthy Eating Index (AHEI, 0-100 points), the Dietary Approach to Stop Hypertension index (DASHi, 8-40 points), the healthy plant-based diet index (hPDI, 18-90 points) and the unhealthy plant-based diet index (uPDI, 18-90 points). substance use will be assessed in a self-reported fashion using a questionnaire.
Relationship between diet quality and alcohol consumption. | Diet questionnaire completion and lifestyle habit measurement will be completed with a 3 weeks period.
  Diet quality indices reflecting different dimensions of diet will be used as the main exposure, including the Alternative Mediterranean Diet Index (AMED, 9-45 points), the Alternative Healthy Eating Index (AHEI, 0-100 points), the Dietary Approach to Stop Hypertension index (DASHi, 8-40 points), the healthy plant-based diet index (hPDI, 18-90 points) and the unhealthy plant-based diet index (uPDI, 18-90 points). Alcohol consumption will be assessed from the food frequency questionnaire.
Relationship between diet quality and medication adherence. | Diet questionnaire completion and lifestyle habit measurement will be completed with a 3 weeks period.
  Diet quality indices reflecting different dimensions of diet will be used as the main exposure, including the Alternative Mediterranean Diet Index (AMED, 9-45 points), the Alternative Healthy Eating Index (AHEI, 0-100 points), the Dietary Approach to Stop Hypertension index (DASHi, 8-40 points), the healthy plant-based diet index (hPDI, 18-90 points) and the unhealthy plant-based diet index (uPDI, 18-90 points). Medication adherence will be assessed using the Medication Adherence Report Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Drouin-Chartier, Study Director — Laval University; Jean-Philippe Drouin-Chartier, Principal Investigator — Laval University
Locations (1):
- Institute of nutrition and functional foods, Laval University, Québec, Canada

IPD SHARING:
Plan to Share IPD: No